CLINICAL TRIAL: NCT01336712
Title: A Phase II Trial of Total Body Irradiation-Based Myeloablative Conditioning and Transplantation of Partially HLA-Mismatched Peripheral Blood Stem Cells for Patients With Hematologic Malignancies
Brief Title: Total Body Irradiation/Fludarabine Based Ablative Haploidentical Transplant for Hematologic Diseases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northside Hospital, Inc. (Other)
Collaborators: Blood and Marrow Transplant Group of Georgia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSH 922
Record Dates: First submitted 2011-04-14; First posted 2011-04-18 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Leukemia; Acute Leukemia; Hodgkin's Disease; Non-Hodgkin's Lymphoma; Myelodysplastic Syndrome
Keywords: CML; CLL; AML; ALL; MDS; HD; NHL; MFB; P.vera; Essential Thrombocytosis
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes; Thrombocythemia, Essential | interventions — Peripheral Blood Stem Cell Transplantation; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Myeloablative Haploidentical Transplant (Experimental): Haplo transplant
  Interventions: Procedure: Peripheral Blood Stem Cell Transplant

INTERVENTIONS:
Procedure: Peripheral Blood Stem Cell Transplant — Total Body Irradiation 1200cGy (150cGy given in 8 fractions twice a day six hours apart on days -4, -3, -2 and -1.
  Fludarabine 30 mg/m^2 given once a day for 3 days on days -7, -6 and -5 Cyclophosphamide 50mg/kg given one a day on days +3 and +4
  Other Names: TBI; Fludara; Cytoxan

SUMMARY:
In this study, patients will receive a myeloablative preparative regimen consisting of fludarabine and total body irradiation (TBI), followed by a T cell replete, mobilized peripheral blood stem cell (PBSC) allograft from a partially matched related donor. All patients will receive post-transplant Cy in addition to standard post transplant immunosuppression with tacrolimus and MMF. The treatment protocol will be essentially identical to the prior study, with the exception of the substitution of TBI for Busulfan. The investigators hypothesize that this change will significantly reduce the risk of HC, while maintaining the efficacy of the transplant.

DETAILED DESCRIPTION:
Historically, haploidentical HSCT has been associated with significant risks of graft rejection and severe graft versus host disease (GVHD), leading to high treatment related mortality and poor outcomes. The risk of engraftment failure and GVHD may be reduced in intensively conditioned recipients of grafts that have been rigorously depleted of T cells, but the risks of serious infection and death from prolonged immune compromise in these patients remains high. Recently, investigators from Johns Hopkins University demonstrated a new approach to haploidentical transplantation, utilizing a nonmyeloablative preparative regimen, followed by a T cell-replete bone marrow infusion and post-transplantation immunosuppression with high dose Cyclophosphamide (Cy), tacrolimus, and MMF. Clinical studies have shown this approach to be safe and effective with a low incidence of graft rejection, GVHD, and treatment-related mortality. Relapse represents the major cause of treatment failure in these patients, particularly with high-risk myeloid malignancies.

In order to decrease this relapse risk in high-risk patients, the investigators initiated a myeloablative haploidentical HSCT study in January 2009 utilizing Busulfan-based conditioning, post-transplant Cy, and PBSC, instead of BM, as the stem cell source. Outcomes of the 15 patients transplanted to date have been promising with 100% engraftment, low rates of treatment-related mortality, relapse and GVHD, and excellent survival rates. An unexpected outcome of the study was a higher-than-expected rate of BK virus-induced hemorrhagic cystitis (HC) occurring in 7 of 14 evaluable patients. Although there were no deaths attributable to HC, it was associated with significant morbidity in some patients.

HC is a recognized complication of allogeneic transplant therapy. Late onset HC, occurring after engraftment, is due almost exclusively to reactivation of the polyoma BK virus (BKV). Other important risk factors associated with HC include Busulfan-based conditioning, acute GVHD, HLA mismatched transplants, and use of bone marrow as the stem cell source. TBI-based conditioning, prior to myeloablative allogeneic transplant, has been associated with significantly less HC than Busulfan-based conditioning in both retrospective and prospective randomized trials.

Eighteen patients will be accrued to this study. The primary end point of this study is the incidence of HC. The investigators will also examine the incidence of acute and chronic GVHD, engraftment, degree of donor-host chimerism, transplant related morbidity and mortality, as well as disease-free and overall survival. Stopping rules will minimize the risk of untoward or unexpected side effects.

ELIGIBILITY:
Inclusion Criteria:

* No available matched related or unrelated donor OR a matched related or unrelated donor that is unavailable in the time frame necessary
* Availability of a 3/6 or 5/6 matched (HLA-A, B, DR) related donor
* Donor must have a negative HLA cross-match in the host vs. graft direction
* Donor must be willing to donate mobilized peripheral blood stem cells
* Age 18 to </=60 years
* Karnofsky Status >/= 70%
* Must have one of the following high-risk malignancies
* Chronic Myelogenous Leukemia (CML) in chronic phase, resistant and/or intolerant to TKI
* CML in accelerated phase
* CML blast crisis that has entered into 2nd Chronic phase following induction
* Acute Myelogenous Leukemia (AML) in 2nd or subsequent complete remission (CR)
* AML primary induction failure but subsequently in CR
* AML in 1st CR with poor risk cytogenetics or arising from preceding hematologic disease
* AML with marrow blasts <5% but persistence of minimal residual disease by flow cytometry, cytogenetics or FISH
* Myelodysplastic Syndrome (MDS) that is treatment related
* MDS that has monosomy 7 or complex cytogenetics
* MDS with IPSS score of 1.5 or greater
* Chronic myelomonocytic leukemia (CMML)
* Acute Lymphocytic Leukemia/lymphoblastic lymphoma (ALL) in 2nd or subsequent complete remission (CR)
* ALL with poor-risk karyotype [t(9;22) or bcr-abl fusion, t(4;11) or other MLL translocation] and in 1st CR
* ALL with marrow blasts < 5% but persistence of minimal residual disease by flow cytometry, cytogenetics or FISH
* Chronic Lymphocytic Leukemia (CLL)/Prolymphocytic Leukemia (PLL) with previously treated disease that has either relapsed or failed to respond adequately to conventional-dose therapy including purine analogs AND in the opinion of the transplant physician is unlikely to benefit from reduced intensity transplantation due to the presence of one or more high risk features (i.e. bulky tumor masses, B symptoms, and/or inadequate response to salvage chemotherapy)
* Hodgkin's or Non-Hodgkin's Lymphoma (including low-grade, mantle cell, and intermediate-grade/diffuse) with previously treated disease that has either relapsed or failed to respond adequately to conventional-dose therapy or autologous transplantation AND in the opinion of the transplant physician is unlikely to benefit from reduced intensity transplantation due to the presence of one or more high risk features (i.e. bulky tumor masses, B symptoms, and/or inadequate response to salvage chemotherapy)
* Advance Myelofibrosis, Primary or Post-Polycythemia Vera/Essential Thrombocythemia. Patients must have one of more of the following accelerate phase features, which have been associated with a median overall survival of </= 15 months
* Blood or bone marrow blasts >/= 10%
* Platelets < 50 x 10*9/L
* Chromosome 17 aberrations

Exclusion Criteria:

* Patients will not be excluded on the basis of sex, racial or ethnic background
* Poor cardiac function: Left ventricular ejection fraction < 45%
* Poor pulmonary function: FEV1 and FVD < 60% predicted
* Poor liver function: bilirubin >/= 2.5 mg/dl (not due to hemolysis, Gilbert's or primary malignancy), AST/ALT > 3x ULN
* Poor renal function: Creatinine >/= 2.0 mg/dl or creatinine clearance (calculated creatinine clearance is permitted) < 40 mL/min based on Traditional Cockcroft-Gault formula: 140-age (yrs) x smaller of actual weight vs ideal body weight (kg)/72 x serum creatinine (mg/dl)
* HIV positive
* Women of childbearing potential who currently are pregnant or who are not practicing adequate contraception
* Patients who have any debilitating medical or psychiatric illness which would preclude their giving informed consent or their receiving optimal treatment and follow-up.
* Prior irradiation therapy rendering patient ineligible for TBI

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott R Solomon, MD, Principal Investigator — Blood and Marrow Transplant Group of Georgia
Locations (1):
- Northside Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Background] Szydlo R, Goldman JM, Klein JP, Gale RP, Ash RC, Bach FH, Bradley BA, Casper JT, Flomenberg N, Gajewski JL, Gluckman E, Henslee-Downey PJ, Hows JM, Jacobsen N, Kolb HJ, Lowenberg B, Masaoka T, Rowlings PA, Sondel PM, van Bekkum DW, van Rood JJ, Vowels MR, Zhang MJ, Horowitz MM. Results of allogeneic bone marrow transplants for leukemia using donors other than HLA-identical siblings. J Clin Oncol. 1997 May;15(5):1767-77. doi: 10.1200/JCO.1997.15.5.1767. PMID 9164184
- [Background] Zuckerman T, Rowe JM. Alternative donor transplantation in acute myeloid leukemia: which source and when? Curr Opin Hematol. 2007 Mar;14(2):152-61. doi: 10.1097/MOH.0b013e328017f64d. PMID 17255793
- [Background] Anasetti C, Amos D, Beatty PG, Appelbaum FR, Bensinger W, Buckner CD, Clift R, Doney K, Martin PJ, Mickelson E, et al. Effect of HLA compatibility on engraftment of bone marrow transplants in patients with leukemia or lymphoma. N Engl J Med. 1989 Jan 26;320(4):197-204. doi: 10.1056/NEJM198901263200401. PMID 2643045
- [Background] Anasetti C, Beatty PG, Storb R, Martin PJ, Mori M, Sanders JE, Thomas ED, Hansen JA. Effect of HLA incompatibility on graft-versus-host disease, relapse, and survival after marrow transplantation for patients with leukemia or lymphoma. Hum Immunol. 1990 Oct;29(2):79-91. doi: 10.1016/0198-8859(90)90071-v. PMID 2249952
- [Background] Kanda Y, Chiba S, Hirai H, Sakamaki H, Iseki T, Kodera Y, Karasuno T, Okamoto S, Hirabayashi N, Iwato K, Maruta A, Fujimori Y, Furukawa T, Mineishi S, Matsuo K, Hamajima N, Imamura M. Allogeneic hematopoietic stem cell transplantation from family members other than HLA-identical siblings over the last decade (1991-2000). Blood. 2003 Aug 15;102(4):1541-7. doi: 10.1182/blood-2003-02-0430. Epub 2003 Apr 24. PMID 12714500
- [Background] Kernan NA, Flomenberg N, Dupont B, O'Reilly RJ. Graft rejection in recipients of T-cell-depleted HLA-nonidentical marrow transplants for leukemia. Identification of host-derived antidonor allocytotoxic T lymphocytes. Transplantation. 1987 Jun;43(6):842-7. PMID 3296349
- [Background] Kernan NA, Collins NH, Juliano L, Cartagena T, Dupont B, O'Reilly RJ. Clonable T lymphocytes in T cell-depleted bone marrow transplants correlate with development of graft-v-host disease. Blood. 1986 Sep;68(3):770-3. PMID 3527302
- [Background] Aversa F, Tabilio A, Velardi A, Cunningham I, Terenzi A, Falzetti F, Ruggeri L, Barbabietola G, Aristei C, Latini P, Reisner Y, Martelli MF. Treatment of high-risk acute leukemia with T-cell-depleted stem cells from related donors with one fully mismatched HLA haplotype. N Engl J Med. 1998 Oct 22;339(17):1186-93. doi: 10.1056/NEJM199810223391702. PMID 9780338
- [Background] Mehta J, Singhal S, Gee AP, Chiang KY, Godder K, Rhee Fv Fv, DeRienzo S, O'Neal W, Lamb L, Henslee-Downey PJ. Bone marrow transplantation from partially HLA-mismatched family donors for acute leukemia: single-center experience of 201 patients. Bone Marrow Transplant. 2004 Feb;33(4):389-96. doi: 10.1038/sj.bmt.1704391. PMID 14716338
- [Background] Aversa F, Terenzi A, Tabilio A, Falzetti F, Carotti A, Ballanti S, Felicini R, Falcinelli F, Velardi A, Ruggeri L, Aloisi T, Saab JP, Santucci A, Perruccio K, Martelli MP, Mecucci C, Reisner Y, Martelli MF. Full haplotype-mismatched hematopoietic stem-cell transplantation: a phase II study in patients with acute leukemia at high risk of relapse. J Clin Oncol. 2005 May 20;23(15):3447-54. doi: 10.1200/JCO.2005.09.117. Epub 2005 Mar 7. PMID 15753458
- [Background] Lang P, Greil J, Bader P, Handgretinger R, Klingebiel T, Schumm M, Schlegel PG, Feuchtinger T, Pfeiffer M, Scheel-Walter H, Fuhrer M, Martin D, Niethammer D. Long-term outcome after haploidentical stem cell transplantation in children. Blood Cells Mol Dis. 2004 Nov-Dec;33(3):281-7. doi: 10.1016/j.bcmd.2004.08.017. PMID 15528145
- [Background] Waller EK, Giver CR, Rosenthal H, Somani J, Langston AA, Lonial S, Roback JD, Li JM, Hossain MS, Redei I. Facilitating T-cell immune reconstitution after haploidentical transplantation in adults. Blood Cells Mol Dis. 2004 Nov-Dec;33(3):233-7. doi: 10.1016/j.bcmd.2004.08.009. PMID 15528137
- [Background] Guinan EC, Boussiotis VA, Neuberg D, Brennan LL, Hirano N, Nadler LM, Gribben JG. Transplantation of anergic histoincompatible bone marrow allografts. N Engl J Med. 1999 Jun 3;340(22):1704-14. doi: 10.1056/NEJM199906033402202. PMID 10352162
- [Background] Rizzieri DA, Koh LP, Long GD, Gasparetto C, Sullivan KM, Horwitz M, Chute J, Smith C, Gong JZ, Lagoo A, Niedzwiecki D, Dowell JM, Waters-Pick B, Liu C, Marshall D, Vredenburgh JJ, Gockerman J, Decastro C, Moore J, Chao NJ. Partially matched, nonmyeloablative allogeneic transplantation: clinical outcomes and immune reconstitution. J Clin Oncol. 2007 Feb 20;25(6):690-7. doi: 10.1200/JCO.2006.07.0953. Epub 2007 Jan 16. PMID 17228020

RESULTS

PARTICIPANT FLOW:
Groups:
- Myeloablative Haploidentical Transplant: Haplo transplant
  Peripheral Blood Stem Cell Transplant: Total Body Irradiation 1200cGy (150cGy given in 8 fractions twice a day six hours apart on days -4, -3, -2 and -1.
  Fludarabine 30 mg/m^2 given once a day for 3 days on days -7, -6 and -5 Cyclophosphamide 50mg/kg given one a day on days +3 and +4
  Patient follow up x6 months
Period: Overall Study
Arm/Group | Myeloablative Haploidentical Transplant
Started | 30
Completed | 27
Not Completed | 3
Not completed — Death | 2
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Groups:
- Myeloablative Haploidentical Transplant: Haplo transplant
  Peripheral Blood Stem Cell Transplant: Total Body Irradiation 1200cGy (150cGy given in 8 fractions twice a day six hours apart on days -4, -3, -2 and -1.
  Fludarabine 30 mg/m2 given once a day for 3 days on days -7, -6 and -5 Cyclophosphamide 50mg/kg given one a day on days +3 and +4
Arm/Group | Myeloablative Haploidentical Transplant
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 13
Race/Ethnicity, Customized [Number; unit: participants]
  White | 10
  Black/African America | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Experiencing Hemorrhagic Cystitis Post Transplant
Description: 1.1 To estimate the incidence of BK virus-associated hemorrhagic cystitis following a TBI-based myeloablative haploidentical HSCT in patients with high risk hematologic malignancies.
Time Frame: 6 months
Measure: Number; unit: percentage of patients
Arm/Group | Myeloablative Haploidentical Transplant
Number analyzed (Participants) | 30
percentage of patients | 30

2. Secondary Outcome: Survival
Description: To obtain estimate of overall survival (OS)
Time Frame: 2 year
Measure: Number; unit: percentage of patients analyzed
Arm/Group | Myeloablative Haploidentical Transplant
Number analyzed (Participants) | 30
percentage of patients analyzed | 78

3. Secondary Outcome: Percentage of Participatns With Donor Chimerism Post-transplant
Description: Characterize donor hematopoietic chimerism in peripheral blood at day 30 after HSCT.
Time Frame: Day 30
Measure: Number; unit: percentage of patients
Arm/Group | Myeloablative Haploidentical Transplant
Number analyzed (Participants) | 30
percentage of patients | 100

4. Secondary Outcome: Disease Free Survival (DFS) Percentage
Time Frame: 2 year
Measure: Number; unit: percentage of patients analyzed
Arm/Group | Myeloablative Haploidentical Transplant
Number analyzed (Participants) | 30
percentage of patients analyzed | 73

5. Secondary Outcome: Non-relapsed Mortality (NRM) Percentage
Time Frame: 2 year
Measure: Number; unit: percentage of patients
Arm/Group | Myeloablative Haploidentical Transplant
Number analyzed (Participants) | 30
percentage of patients | 3

6. Secondary Outcome: Relapse Rate
Time Frame: 2 year
Measure: Number; unit: percentage of patients analyzed
Arm/Group | Myeloablative Haploidentical Transplant
Number analyzed (Participants) | 30
percentage of patients analyzed | 24

7. Secondary Outcome: Cumulative Incidence of Chronic Graft-versus-host Disease
Time Frame: 2 year
Measure: Number; unit: percentage of patients analyzed
Arm/Group | Myeloablative Haploidentical Transplant
Number analyzed (Participants) | 30
percentage of patients analyzed | 56

ADVERSE EVENTS:
Arm/Group | Myeloablative Haploidentical Transplant
Serious Adverse Events (participants affected / at risk) | 13/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myeloablative Haploidentical Transplant (N=30)
Veno-Occlusive Disease (Hepatobiliary disorders) | 1 (1)
BK Virus (Infections and infestations) | 1 (1)
anorexia (Gastrointestinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hemolytic Uremic Syndrom (Blood and lymphatic system disorders) | 1 (1)
Nausea & vomiting (Gastrointestinal disorders) | 1 (1)
Renal Insufficiency (Renal and urinary disorders) | 2 (2)
Alveolar Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Syncope (Cardiac disorders) | 1 (1)
Sepsis syndrome (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myeloablative Haploidentical Transplant (N=30)
abcessed tooth (Gastrointestinal disorders) | 2 (2)
abdominal bloating (Gastrointestinal disorders) | 6 (6)
abdominal cramping/discomfort (Gastrointestinal disorders) | 20 (20)
abdominal fullness (Gastrointestinal disorders) | 2 (2)
abdominal muscle soreness (secondary to cough) (Gastrointestinal disorders) | 2 (2)
abdominal tenderness (Gastrointestinal disorders) | 8 (8)
abnormal gait (Nervous system disorders) | 2 (2)
acidosis (Gastrointestinal disorders) | 4 (4)
acute GVHD - gut (Immune system disorders) | 10 (10)
acute GVHD - skin (Immune system disorders) | 8 (8)
agitation (Psychiatric disorders) | 2 (2)
increased alkaline phosphatase (Hepatobiliary disorders) | 20 (20)
increased ALT (Hepatobiliary disorders) | 22 (22)
neutropenia (Blood and lymphatic system disorders) | 26 (26)
anorexia (Gastrointestinal disorders) | 15 (15)
anxiety (Psychiatric disorders) | 26 (26)
increased AST (Hepatobiliary disorders) | 29 (29)
atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
BK Virus (Renal and urinary disorders) | 10 (10)
bladder mass (Renal and urinary disorders) | 2 (2)
bladder pressure (Renal and urinary disorders) | 2 (2)
bladder spasms (Renal and urinary disorders) | 3 (3)
bleeding gums (Blood and lymphatic system disorders) | 5 (5)
blood clots in urine (Renal and urinary disorders) | 2 (2)
blood in sputum (Blood and lymphatic system disorders) | 2 (2)
blurred vision (Nervous system disorders) | 7 (7)
benign prostatic hyperplasia (Renal and urinary disorders) | 3 (3)
bradycardia (Cardiac disorders) | 6 (6)
bruising (Blood and lymphatic system disorders) | 6 (6)
bumps on skin (Skin and subcutaneous tissue disorders) | 2 (2)
c.difficile colitis (Infections and infestations) | 5 (5)
chest discomfort with inspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
chest tightness (Cardiac disorders) | 2 (2)
chills (Investigations) | 22 (22)
CMV reactivation (Blood and lymphatic system disorders) | 15 (15)
coarse breath sounds (Respiratory, thoracic and mediastinal disorders) | 6 (6)
coated tongue (Gastrointestinal disorders) | 5 (5)
confusion (Nervous system disorders) | 2 (2)
constipation (Gastrointestinal disorders) | 19 (19)
dry cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
cough NOS (Respiratory, thoracic and mediastinal disorders) | 21 (21)
increased creatinine (Renal and urinary disorders) | 16 (16)
CVC site bleeding (Investigations) | 2 (2)
CVC site edema (Investigations) | 2 (2)
CVC site soreness (Investigations) | 3 (3)
CVC site tenderness (Investigations) | 7 (7)
deconditioned (Investigations) | 20 (20)
decreased appetite (Gastrointestinal disorders) | 22 (22)
decreased breath sounds (Respiratory, thoracic and mediastinal disorders) | 15 (15)
decreased fluid intake (Gastrointestinal disorders) | 7 (7)
decreased oral intake (Gastrointestinal disorders) | 5 (5)
dehydration (Investigations) | 5 (5)
depression (Psychiatric disorders) | 19 (19)
diaphoresis (Skin and subcutaneous tissue disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 30 (30)
difficulty swallowing (Gastrointestinal disorders) | 10 (10)
labored breathing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
abdominal distention (Gastrointestinal disorders) | 8 (8)
dizziness (Nervous system disorders) | 16 (16)
drowsiness (Nervous system disorders) | 18 (18)
dry heaves (Gastrointestinal disorders) | 5 (5)
dry lips (Gastrointestinal disorders) | 3 (3)
dry mouth (Gastrointestinal disorders) | 18 (18)
dry skin (Skin and subcutaneous tissue disorders) | 19 (19)
dry throat (Gastrointestinal disorders) | 3 (3)
dysgeusia (Gastrointestinal disorders) | 5 (5)
dyspepsia (Gastrointestinal disorders) | 2 (2)
dysphagia (Gastrointestinal disorders) | 6 (6)
dysuria (Renal and urinary disorders) | 18 (18)
ear fullness (Ear and labyrinth disorders) | 2 (2)
edema of hands and feet (Cardiac disorders) | 2 (2)
lower extremity edema (Cardiac disorders) | 18 (18)
electrolyte wasting syndrome (Metabolism and nutrition disorders) | 6 (6)
epistaxis (Blood and lymphatic system disorders) | 11 (11)
generalized erythema (Skin and subcutaneous tissue disorders) | 7 (7)
throat erythema (Skin and subcutaneous tissue disorders) | 3 (3)
erythematous palms (Skin and subcutaneous tissue disorders) | 2 (2)
esophagitis (Gastrointestinal disorders) | 9 (9)
esophageal pain (Gastrointestinal disorders) | 3 (3)
exertional shortness of breath (Respiratory, thoracic and mediastinal disorders) | 5 (5)
facial flushing (Skin and subcutaneous tissue disorders) | 4 (4)
fatigue (Investigations) | 29 (29)
fever (Investigations) | 24 (24)
left lower flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
flat affect (Psychiatric disorders) | 11 (11)
flatulence (Gastrointestinal disorders) | 3 (3)
fluid overload (Cardiac disorders) | 11 (11)
folliculitis (Infections and infestations) | 4 (4)
gastritis (Gastrointestinal disorders) | 3 (3)
generalized body aches (Musculoskeletal and connective tissue disorders) | 11 (11)
GERD (Gastrointestinal disorders) | 24 (24)
gastrointenstinal bleed (Gastrointestinal disorders) | 2 (2)
hallucinations (Psychiatric disorders) | 2 (2)
headache (Nervous system disorders) | 24 (24)
hematuria (Renal and urinary disorders) | 11 (11)
hemoptysis (Blood and lymphatic system disorders) | 2 (2)
hemorrhoids (Gastrointestinal disorders) | 5 (5)
anemia (Blood and lymphatic system disorders) | 28 (28)
hiccups (Gastrointestinal disorders) | 4 (4)
hyperactive bowel sounds (Gastrointestinal disorders) | 3 (3)
hyperbilirubinemia (Hepatobiliary disorders) | 8 (8)
hypercalcemia (Metabolism and nutrition disorders) | 10 (10)
hyperglycemia (Metabolism and nutrition disorders) | 30 (30)
hyperkalemia (Metabolism and nutrition disorders) | 15 (15)
hypermagnesemia (Metabolism and nutrition disorders) | 3 (3)
hypernatremia (Metabolism and nutrition disorders) | 19 (19)
hyperpigmented skin (Skin and subcutaneous tissue disorders) | 13 (13)
hypertension (Cardiac disorders) | 27 (27)
hypoactive bowel sounds (Gastrointestinal disorders) | 5 (5)
hypoalbuminemia (Metabolism and nutrition disorders) | 24 (24)
hypocalcemia (Metabolism and nutrition disorders) | 25 (25)
hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
hypokalemia (Metabolism and nutrition disorders) | 23 (23)
hypomagnesemia (Metabolism and nutrition disorders) | 27 (27)
hyponatremia (Metabolism and nutrition disorders) | 10 (10)
hypotension (Cardiac disorders) | 19 (19)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
stool incontinence (Gastrointestinal disorders) | 7 (7)
bacteremia infection (NOS) (Infections and infestations) | 6 (6)
influenza (Infections and infestations) | 2 (2)
insomnia (Psychiatric disorders) | 23 (23)
irregular heartbeat (Cardiac disorders) | 4 (4)
leg cramping (Musculoskeletal and connective tissue disorders) | 5 (5)
leg discomfort (2nd lower extremity edema) (Musculoskeletal and connective tissue disorders) | 2 (2)
lethargy (Investigations) | 11 (11)
lightheadedness (Nervous system disorders) | 3 (3)
limited mobility (Musculoskeletal and connective tissue disorders) | 9 (9)
limited sensory perception (Nervous system disorders) | 6 (6)
loss of balance (Nervous system disorders) | 8 (8)
lower extremity pain (Musculoskeletal and connective tissue disorders) | 3 (3)
lung crackles (Respiratory, thoracic and mediastinal disorders) | 7 (7)
lung infiltrates (Respiratory, thoracic and mediastinal disorders) | 4 (4)
lymphocytopenia (Blood and lymphatic system disorders) | 12 (12)
malaise (Investigations) | 7 (7)
malnutrition (Gastrointestinal disorders) | 2 (2)
melena (Gastrointestinal disorders) | 2 (2)
menstrual cramps (Reproductive system and breast disorders) | 3 (3)
metapneumovirus (Respiratory, thoracic and mediastinal disorders) | 2 (2)
migraine headaches (Nervous system disorders) | 3 (3)
mouth sores (Gastrointestinal disorders) | 10 (10)
mucositis (Gastrointestinal disorders) | 25 (25)
myalgias (Musculoskeletal and connective tissue disorders) | 2 (2)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 (9)
nausea (Gastrointestinal disorders) | 29 (29)
febrile neutropenia (Blood and lymphatic system disorders) | 26 (26)
night sweats (Investigations) | 3 (3)
nocturia (Renal and urinary disorders) | 3 (3)
oral candida (Infections and infestations) | 2 (2)
oral lesions (Gastrointestinal disorders) | 2 (2)
oral thrush (Investigations) | 10 (10)
orthostatic hypotension (Cardiac disorders) | 3 (3)
abdominal pain (Gastrointestinal disorders) | 13 (13)
ankle pain (Musculoskeletal and connective tissue disorders) | 3 (3)
arm pain (Musculoskeletal and connective tissue disorders) | 3 (3)
back pain (Musculoskeletal and connective tissue disorders) | 10 (10)
bladder pain (Renal and urinary disorders) | 2 (2)
bone pain (Musculoskeletal and connective tissue disorders) | 4 (4)
chest pain (Musculoskeletal and connective tissue disorders) | 6 (6)
chest pain (2nd cough) (Musculoskeletal and connective tissue disorders) | 3 (3)
CVC site pain (Investigations) | 3 (3)
fingertip pain (Musculoskeletal and connective tissue disorders) | 2 (2)
foot pain (Musculoskeletal and connective tissue disorders) | 5 (5)
hand pain (Musculoskeletal and connective tissue disorders) | 6 (6)
hemorrhoidal pain (Gastrointestinal disorders) | 2 (2)
jaw pain (Musculoskeletal and connective tissue disorders) | 4 (4)
joint pain (Musculoskeletal and connective tissue disorders) | 8 (8)
knee pain (Musculoskeletal and connective tissue disorders) | 4 (4)
leg pain (Musculoskeletal and connective tissue disorders) | 10 (10)
mouth pain (Gastrointestinal disorders) | 13 (13)
muscle pain (Musculoskeletal and connective tissue disorders) | 3 (3)
shoulder pain (Musculoskeletal and connective tissue disorders) | 4 (4)
throat pain (2nd mucositis) (Gastrointestinal disorders) | 5 (5)
tooth pain (Gastrointestinal disorders) | 2 (2)
pain with swallowing (Gastrointestinal disorders) | 4 (4)
pale skin (Skin and subcutaneous tissue disorders) | 2 (2)
palpitations (Cardiac disorders) | 4 (4)
panic attack (Nervous system disorders) | 2 (2)
parainfluenza (Infections and infestations) | 2 (2)
parotid gland edema (Investigations) | 2 (2)
parotid gland tenderness (Investigations) | 2 (2)
parotitis (Infections and infestations) | 2 (2)
pericardial effusion (Cardiac disorders) | 3 (3)
peripheral neuropathy (Nervous system disorders) | 16 (16)
perirectal irritation (Gastrointestinal disorders) | 5 (5)
perirectal pain (Gastrointestinal disorders) | 3 (3)
petechiae (Blood and lymphatic system disorders) | 5 (5)
photosensitivity (Nervous system disorders) | 2 (2)
platelet infusion reaction (Investigations) | 2 (2)
thrombocytopenia (Blood and lymphatic system disorders) | 29 (29)
pneumonia (Infections and infestations) | 4 (4)
postnasal drainage (Respiratory, thoracic and mediastinal disorders) | 8 (8)
prolonged urine stream (Renal and urinary disorders) | 2 (2)
pruritus (Skin and subcutaneous tissue disorders) | 26 (26)
rales (Respiratory, thoracic and mediastinal disorders) | 4 (4)
rash (Skin and subcutaneous tissue disorders) | 17 (17)
rash (arms, thighs) (Skin and subcutaneous tissue disorders) | 2 (2)
renal failure (Renal and urinary disorders) | 2 (2)
acute renal insufficiency (Renal and urinary disorders) | 13 (13)
respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 4 (4)
restless legs (Nervous system disorders) | 2 (2)
rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 12 (12)
rhinovirus (Infections and infestations) | 2 (2)
rhonchi (Respiratory, thoracic and mediastinal disorders) | 5 (5)
rigors (General disorders) | 6 (6)
saliva thickening (Gastrointestinal disorders) | 3 (3)
scalloped tongue border (Gastrointestinal disorders) | 7 (7)
scrotal edema (Reproductive system and breast disorders) | 2 (2)
seasonal allergies (General disorders) | 6 (6)
sedation (Nervous system disorders) | 3 (3)
serous otitis (Ear and labyrinth disorders) | 2 (2)
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 9 (9)
sinus drainage (Respiratory, thoracic and mediastinal disorders) | 3 (3)
sinus headache (Nervous system disorders) | 2 (2)
sinus pressure (General disorders) | 2 (2)
sinus tenderness (General disorders) | 3 (3)
sinusitis (General disorders) | 5 (5)
skin dyspigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
skin irriation (Skin and subcutaneous tissue disorders) | 2 (2)
skin lesions (Skin and subcutaneous tissue disorders) | 3 (3)
skin tenderness (Skin and subcutaneous tissue disorders) | 3 (3)
small bowel obstruction (Gastrointestinal disorders) | 2 (2)
sneezing (General disorders) | 4 (4)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 14 (14)
somnolence (Nervous system disorders) | 3 (3)
sore throat (Gastrointestinal disorders) | 18 (18)
splenomegaly (Endocrine disorders) | 2 (2)
staphylococcus hemolyticus bacteremia (Infections and infestations) | 2 (2)
steroid-induced diabetes (Metabolism and nutrition disorders) | 3 (3)
stomatitis (Gastrointestinal disorders) | 9 (9)
suprapubic tenderness (Musculoskeletal and connective tissue disorders) | 2 (2)
facial swelling (General disorders) | 2 (2)
tachycardia (Cardiac disorders) | 25 (25)
tachypnea (Cardiac disorders) | 3 (3)
taste alteration (Nervous system disorders) | 10 (10)
thick oral secretions (Gastrointestinal disorders) | 2 (2)
throat swelling (General disorders) | 2 (2)
tongue ridging (Gastrointestinal disorders) | 3 (3)
tongue swelling (General disorders) | 2 (2)
tremors (Nervous system disorders) | 9 (9)
tremors (hands) (Nervous system disorders) | 2 (2)
unsteady gait (Nervous system disorders) | 2 (2)
urinary frequency (Renal and urinary disorders) | 23 (23)
urinary hesitancy (Renal and urinary disorders) | 5 (5)
urinary incontinence (Renal and urinary disorders) | 6 (6)
urinary retention (Renal and urinary disorders) | 4 (4)
urinary urgency (Renal and urinary disorders) | 16 (16)
vaginal bleeding/spotting (Reproductive system and breast disorders) | 7 (7)
volume depletion (General disorders) | 6 (6)
volume overload (General disorders) | 3 (3)
vomiting (Gastrointestinal disorders) | 24 (24)
vancomycin-resistant enterococci (Infections and infestations) | 5 (5)
leukopenia (Blood and lymphatic system disorders) | 28 (28)
weakness (General disorders) | 24 (24)
weight gain (Gastrointestinal disorders) | 3 (3)
weight loss (Gastrointestinal disorders) | 22 (22)
wheezing (Respiratory, thoracic and mediastinal disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No